CLINICAL TRIAL: NCT00643721
Title: Body Water Content Sensor
Status: Terminated | Type: Observational
Why Stopped: Record owner left institution
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Lori Ploutz-Snyder, Syracuse University
Other Study IDs: 5408
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Young healthy athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- D,FR: Young healthy athletes
  Interventions: Other: dehydration

INTERVENTIONS:
Other: dehydration — dehydration to 3% and 5% loss of total body water

SUMMARY:
Evaluation of hydration status during exercise and heat exposure.

DETAILED DESCRIPTION:
Evaluation of hydration status during exercise and heat exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Participates in regular exercise
* Able to tolerate exercise in the heat

Exclusion Criteria:

* Abnormal hemoglobin
* Any exercise limitations
* Pregnancy
* Cardiovascular or orthopedic disease/conditions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy athletes
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Body weight and hydration status | Before exercise and following dehydration

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Human Performance, Syracuse, New York, United States